CLINICAL TRIAL: NCT03700697
Title: A Clinical Process Support System for Primary Care to Address Family Stress
Acronym: FamilyStress
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Total Child Health, Inc. (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Center for Promotion of Child Development through Primary Care (Unknown); Foresight Logic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R44HD089785 (NIH); R44HD089785 (NIH)
Record Dates: First submitted 2018-07-14; First posted 2018-10-09 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Social Determinants of Health; Child Abuse

STUDY DESIGN:
Intervention Model Description: A cluster randomized quality improvement intervention trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Stress Module Intervention (Experimental): Primary care clinicians will use the CHADIS Family Stress Module including the reviewing ACE, Positive Childhood Experiences, and FASS Plus questionnaires at designated child ages; address family stressors revealed using the motivational interviewing teleprompter and refer parents with stressors as indicated using the care coordination functionality.
  Interventions: Behavioral: Family Stress Module Intervention
- Controls (No Intervention): Control primary care providers will provide care as usual.

INTERVENTIONS:
Behavioral: Family Stress Module Intervention — as above
  Arms: Family Stress Module Intervention

SUMMARY:
This project is to create and test a "clinical process support system" that will improve the ability of primary child health care providers (PCPs) to screen for and address family stressors during routine child health visits that are associated with negative child outcomes in a manner that is feasible and acceptable to both clinicians and parents.

DETAILED DESCRIPTION:
This project is to create and test a "clinical process support system" that will improve the ability of primary child health care providers (PCPs) to screen for and address family stressors during routine child health visits that are associated with negative child outcomes in a manner that is feasible and acceptable to both clinicians and parents. The family stressors assessed include: intimate partner violence (IPV), parental depression, parental stress, food insecurity, parental substance use and harsh punishment of the child. The system is designed to overcome known obstacles to addressing these issues during routine well child visits. These obstacles include: lack of PCP training in an evidence-based approach to the interview (e.g., motivational interviewing); lack of time; low parental expectations for addressing sensitive family issues during routine child "physicals"; and the usual absence of co-located mental health providers. The new Family Stress module will build on two foundations: 1) previous studies of screening using the Safe Environment for Every Kid (SEEK) tool, which showed reduced child maltreatment outcomes in two Randomized Control Trials; and 2) an existing online screening and decision support system (CHADIS). The goals are to support parents in reducing family risk and the exposure of the young child to their own Adverse Childhood Experiences (ACE), including child maltreatment.

The innovations in this method of addressing family stressors and overcoming the above obstacles include:

1. Time efficiencies. Time is saved through pre-visit online data collection, saving both interview and clinical documentation time and staff time saved for patient education and needed referrals.
2. Creating the environment for psychosocial care. This is done through a combination of pre-visit questionnaires with agenda broadening questions (best and hardest parts of parenting), inclusion of parental background from Adverse Childhood Experiences (ACE) and Positive Childhood Experiences inquiries in clinical discussions; individualized text and resources for the family in the Care Portal; milestones to "celebrate" in each child's "MemoryBook"; and empathetic and reflective responses from the PCP.
3. Efficient training. Training is done using innovative "moment of care" teleprompters created instantly in response to the individual parent issues from the pre-visit tools to support the difficult conversations and a motivational interview begun by the computer needed to move families towards services.
4. Care communication. Practices will be able to share data with their own colocated services or be linked electronically with outside local resources using a unique online "consent to share information" functionality that also facilitates determining if the referral appointment was completed. Visit notes and documentation of attendance at a consultation will be shared with consent between the PCP and referral agency or professional to facilitate two-way communication for coordinated care.

Design: A cluster randomized quality improvement intervention using the clinical process support family stress module in routine care for children 0-3 years will be conducted in 30 primary care practices. The project will enroll as many 0-4 month olds as possible and follow them to age 24 months and a cohort of 18-24 month olds as controls using online consent (not requiring staff time). For this 2.5 year project the study staff will ask physicians and office staff to complete a one hour online training, offices to notify parents to complete CHADIS when scheduling well-child visits for children 0-3 years old with the questionnaire assignments for the project including Family Assessment of Safety and Stress (FASS), and primary care clinicians to use the CHADIS Family Stress module including the care coordination functionality during the visits when that site is randomized to the intervention period. At the end of the project the study requires clinicians to complete a survey and provide information from the medical records for participating children about immunization completion and missed visits. This information can be collected in a variety of ways depending on each electronic record.

Outcomes: The outcomes anticipated for the proposed study include improved parent connection to services and parent-child relationships, and reduced family stressors, child behavior problems, harsh punishment, and Child Protection referrals for abuse and neglect. Expected outcomes include that higher parent satisfaction with the enhanced clinical process will result in lower rates of missed visits and delayed immunizations. These results should provide evidence of the effectiveness of PCP screening and referral to reduce family stressors and the evidence needed for full United States Preventive Services Task Force endorsement of this clinical process support tool for reducing child maltreatment.

ELIGIBILITY:
Inclusion Criteria:

* Parents and their children 1 month to 4 months at enrollment.
* Parents and their children 16-20 months for comparison group.
* Primary Care Providers of any age.

Exclusion Criteria:

-Unable to speak and read English.

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16630 (Estimated)
Dates: Start 2018-07-09 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Compare intervention vs control percent parents for receiving help for Family Stressors | first 2 years of life
  Compare intervention vs control percent parents endorsing "getting help" with any of:
  * Intimate Partner Violence per Hurt, insulted, Threatened with Harm, Screamed score >=2 (0-40)
  * substance use per NIH measure of excess alcohol or drug use >2 (0-12)
  * depression per Patient Health Questionnaire-2 >=2 (0-4),
  * food insecurity per Hunger Vital Sign >=1 (0-2),
  * life stress per parent report of life stress (yes/no)
  * harsh punishment per by report of hitting or screaming >=1(0-2)
Compare intervention vs control percent parents in rates of child maltreatment | first 2 years of life
  Compare difference between groups in percent with allegations of child maltreatment per state Child Protective Services agency.
Compare intervention vs control percent parents in rates of harsh punishment | first 2 years of life
  Compare intervention vs control percent parents for difference between groups in percent with harsh punishment per Conflict Tactics Scale- Parent Child version >0 (0-2)
Compare intervention vs control parents in percent reporting child behavior problems | first 2 years of life
  Compare intervention vs control parents in percent reporting behavior problems per Early Childhood Screening Assessment-short form >=9 (0-44)
Compare intervention vs control percent parents for rate of atypical child development. | first 2 years of life
  Compare intervention vs control parents in rates of atypical child development as measured by Age & Stages Questionnaire (monitoring zone or referral zone are atypical)

SECONDARY OUTCOMES:
Compare parent rating of physician competence and confidence handling family stressors between intervention and control groups | 12 months of child's age (Parent)
  Compare rating total scores of self reported care and confidence on survey measure using vignettes called Patient View of Healthcare.
Change in physician competence and confidence handling family stressors | 2 years from first measure (PCP)
  Change in total score of ratings of self reported care and confidence on survey measure using vignettes at start and end of project, approximately 2.5 years.
Compare intervention vs control group rates of missed well child visits | at 2 years of age
  Difference between groups in percent of medical record reports of missed well child visits (0-6 visits)
Compare intervention vs control group rates of missed recommended immunizations | at 2 years of age
  Difference between groups in percent of medical record reports of missed recommended routine vaccinations (0-5 episodes)
Compare intervention vs control group parent-child relationship | 18 months of age
  Difference between groups on total score on Protective Factors Survey of parent ratings of family relationships (0-140)
Compare intervention vs control group parent-child relationship | 24 months of age
  Difference between groups on total score on Protective Factors Survey of parent ratings of family relationships (0-140)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Howard, MD, Principal Investigator — Total Child Health; Raymond Sturner, MD, Principal Investigator — Ctr for Promotion of Child Dev. through Primary Care
Locations (1):
- Total Child Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Only deidentified data will be available to share. All data will be available to researchers with appropriate interest by arrangement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After study completion and reporting to NIH.
Access Criteria: Researchers with appropriate interest, by arrangement.

DOCUMENTS (1):
  • Informed Consent Form (2019-07-31): https://cdn.clinicaltrials.gov/large-docs/97/NCT03700697/ICF_000.pdf